CLINICAL TRIAL: NCT01317563
Title: Phase 2 Study of Antioxidant Therapy in Lean and Obese Asthmatics
Brief Title: Antioxidant Therapy in Lean and Obese Asthmatics
Acronym: ALOA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Principal Investigator, Jason Lang, PI, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALASE08140ALOA
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: asthma; obesity; nutrition; antioxidant
MeSH Terms: conditions — Asthma; Obesity | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antioxidant arm (Active Comparator): Two capsules twice daily (total daily dose = Vitamin A 10000 IU, Vitamin C 1200mg, Vitamin E 400 IU, Selenium 300mcg)
  Interventions: Dietary Supplement: Vitamins A, E, C & Selenium
- Placebo arm (Placebo Comparator): two capsules twice daily (total daily dose = 1200mg whey protein, 800mg microcrystalline cellulose)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamins A, E, C & Selenium — daily dose = Vitamin A 10000 IU (beta carotene), Vitamin E 400 IU, Vitamin C 1200mg, and Selenium 300mcg.
  Arms: Antioxidant arm
Dietary Supplement: Placebo — total daily dose = 1200mg whey protein, 800mg microcrystalline cellulose
  Arms: Placebo arm

SUMMARY:
This project will assess the effectiveness of antioxidant supplementation with common vitamins A, C, E and selenium in controlling asthma symptoms among lean and obese asthmatics. This project may improve our ability to treat asthma and our understanding of the link between nutritional antioxidants and asthma.

DETAILED DESCRIPTION:
Asthma & Obesity are both growing public health crises that also may be critically interrelated for many patients. Obesity increases the risk for asthma in both adults and children, and obesity increases the severity of existing asthma. Obesity leads to increased systemic oxidative stress, however little is know about obesity-related oxidative stress within the airway. Since oxidative stress contributes to the pathogenesis of asthma, obesity may influence asthma risk and severity through this mechanism. Asthmatics have low serum antioxidant activity. There is conflicting evidence about whether or not antioxidant supplementation reduces asthma severity. This may be related to asthma's heterogeneous nature. Antioxidant supplementation may be effective in select subgroups that have the greater oxidative stress, such as asthmatics with occupational exposures or obesity. In fact, the evidence supporting antioxidant supplementation in asthma involved subjects with oxidant-related triggers. We hypothesize that obesity-related oxidant stress puts asthmatics at risk for increased airway oxidative stress and greater asthma severity. We hypothesize that supplementation with common antioxidants will significantly reduce airway inflammation and oxidative stress, and lead to improved pulmonary function and daily asthma control. This pilot study is designed as a randomized, double-blinded, placebo-controlled, parallel intervention trial involving lean and obese adolescents and young adults with asthma. After the 2-week run-in period, all subjects will undergo baseline testing (see figure 1). At randomization they will receive either placebo or a multivitamin antioxidant for 42 days. At the end of the 42 day intervention all subjects will undergo final testing. Primary Hypothesis: In young asthmatics, antioxidant supplementation increases plasma and airway antioxidant levels leading to improved lung function and asthma control. Secondary Hypotheses: 1) Obesity-related systemic oxidant stress is associated with increased oxidative stress within the airway. 2) Antioxidant supplementation will lead to greater improvements in asthma control among obese compared to lean (not underweight) asthmatics. 3) Antioxidant supplementation will lead to greater improvements in airway markers of inflammation and oxidative stress among obese compared to lean asthmatics. We will assess asthma control and lung function before and after therapy.

ELIGIBILITY:
Inclusion Criteria:

* age 12-25,
* physician-diagnosed persistent asthma on daily controller therapy,
* FEV1% >= 60% predicted,
* Lung responsiveness (>= 12% BD reversibility or PC20 MCT <= 16mg/ml)

Exclusion Criteria:

* taking daily MVI,
* chronic oral steroid therapy,
* BMI<20th percentile,
* smoking history,
* pregnancy,
* milk allergy,
* celiac disease

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2008-07; Primary Completion 2012-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Asthma Control Questionnaire (Juniper)- (ACQ) | 6 weeks
  ACQ is a 7 component test that includes 6 responses elliciting control of asthma symptoms plus one component based on FEV1 (spirometry). The score ranges from 0-6, with a higher score suggesting greater asthma symptoms.

SECONDARY OUTCOMES:
Change in Asthma Symptom Utility Index | 6 weeks
  Questionnaire assessing patient reported asthma symptoms from the previous 2 weeks. Score ranges from 0 to 1 with a higher score suggesting better asthma control.
change in FEV1 | 6 weeks
  Spirometric measure of volume expired in 1 second.

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Lang, M.D., Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States